CLINICAL TRIAL: NCT02541591
Title: Neuroprotective Goal Directed Hemodynamic Optimization in Post-cardiac Arrest Patients: a Randomized Controlled Trial (the NEUROPROTECT Post-CA Trial)
Brief Title: Neuroprotective Goal Directed Hemodynamic Optimization in Post-cardiac Arrest Patients
Acronym: NEUROPROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s58017
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Ischemia; Cardiac Arrest
Keywords: post cardiac arrest; hemodynamics
MeSH Terms: conditions — Brain Ischemia; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuroprotect (Experimental): MAP between 85-100mmHg SVO2 between 65-75%
  Interventions: Other: Neuroprotective goal directed hemodynamic optimization
- Control (Active Comparator): MAP>65mmHg
  Interventions: Other: MAP > 65mmHg

INTERVENTIONS:
Other: Neuroprotective goal directed hemodynamic optimization
  Arms: Neuroprotect
Other: MAP > 65mmHg — MAP > 65mmHg
  Arms: Control

SUMMARY:
The primary objective of the Neuroprotect trial is to assess whether or not a new goal directed hemodynamic optimization strategy can reduce cerebral ischemia in post-cardiac arrest (CA) patients.

DETAILED DESCRIPTION:
Unconscious patients admitted to the intensive care unit after being successfully resuscitated from cardiac arrest (CA) are at high risk for death, and neurological deficits are common among survivors. Nevertheless, the optimal hemodynamic strategy to ensure optimal cerebral perfusion and maximal outcome has not been studied by a randomized controlled trial. In the absence of good evidence, current post-CA guidelines are adapted from sepsis guidelines and recommend targeting a mean arterial pressure (MAP) above 65 mmHg (Peberdy ea, Circulation 2010). Importantly, post-CA patients have a large cerebral penumbra at risk for infarction when resuscitated to suboptimal MAP's. In a large subset of post-CA patients the lower threshold of cerebral autoregulation is shifted rightward and these patients might benefit from resuscitation to higher MAP's (Sundgreen ea, Stroke 2001) in order to ensure adequate cerebral oxygenation. Our research group previously showed that a MAP of 85-100mmHg results in optimal cerebral perfusion in post-CA patients (Ameloot ea, resuscitation 2015). Two retrospective and 2 prospective observational studies suggested an association between higher MAP's and better outcome in post-CA patients (Ameloot ea, resuscitation 2015). However, the value of these trials is limited by their observational design. The question remains as to whether patients with higher MAP's do have a better outcome due to more optimal cerebral perfusion and less cerebral damage or whether a higher MAP is merely a non-causal marker of more limited disease severity in these patients. In other words, the primary research question is whether we can reduce cerebral ischemia and improve prognosis of post-cardiac arrest survivors by targeting higher mean systemic blood pressures thereby optimizing cerebral perfusion during their stay in the intensive care unit. To answer this, we propose a multicenter interventional open label investigator driven randomized controlled trial to compare a goal-directed potentially neuro-protective hemodynamic optimization strategy with the current standard of care. Primary efficacy endpoints of the study will include extent of cerebral damage as assessed with diffusion weighted magnetic resonance imaging (DW-MRI), functional and neurocognitive testing, biomarkers of brain injury and survival rates. The final utilization goal of the Neuroprotect post-CA trial is to show that our adapted hemodynamic protocol reduces cerebral ischemia, and improves survival and functional outcome of post-cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital CA of presumed cardiac cause irrespective of the presenting rhythm
2. Unconsciousness (Glasgow coma scale < 8) at hospital admission
3. Age ≥ 18 years
4. Sustained return of spontaneous circulation (ROSC) (=when chest compressions have not been required for 20 consecutive minutes)

Exclusion Criteria:

1. Suspected or confirmed intracranial bleeding or stroke
2. Known limitations in therapy or Do Not Resuscitate-order
3. Known disease compromising 180 day survival
4. Known pre-CA cerebral performance category 3-4
5. Previous stroke (TIA can be included)
6. MRI incompatible cardiac or neurosurgical device
7. Systolic blood pressure < 90 mmHg on norepinephrine > 1 mcg/kg/min).
8. Open chest
9. ECMO (extracorporeal membrane oxygenation)
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Ameloot, MD, Principal Investigator — UZ Leuven; Stefan Janssens, MD, Principal Investigator — UZ Leuven; Joseph Dens, MD, Principal Investigator — Ziekenhuis Oost-Limburg; Cathy De Deyne, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - UZ Leuven, Leuven

REFERENCES:
- [Derived] Laurikkala J, Ameloot K, Reinikainen M, Palmers PJ, De Deyne C, Bert F, Dupont M, Janssens S, Dens J, Hastbacka J, Jakkula P, Loisa P, Birkelund T, Wilkman E, Vaara ST, Skrifvars MB. The effect of higher or lower mean arterial pressure on kidney function after cardiac arrest: a post hoc analysis of the COMACARE and NEUROPROTECT trials. Ann Intensive Care. 2023 Nov 21;13(1):113. doi: 10.1186/s13613-023-01210-0. PMID 37987871
- [Derived] Wouters A, Scheldeman L, Plessers S, Peeters R, Cappelle S, Demaerel P, Van Paesschen W, Ferdinande B, Dupont M, Dens J, Janssens S, Ameloot K, Lemmens R. Added Value of Quantitative Apparent Diffusion Coefficient Values for Neuroprognostication After Cardiac Arrest. Neurology. 2021 May 25;96(21):e2611-e2618. doi: 10.1212/WNL.0000000000011991. Epub 2021 Apr 9. PMID 33837117
- [Derived] Ameloot K, Jakkula P, Hastbacka J, Reinikainen M, Pettila V, Loisa P, Tiainen M, Bendel S, Birkelund T, Belmans A, Palmers PJ, Bogaerts E, Lemmens R, De Deyne C, Ferdinande B, Dupont M, Janssens S, Dens J, Skrifvars MB. Optimum Blood Pressure in Patients With Shock After Acute Myocardial Infarction and Cardiac Arrest. J Am Coll Cardiol. 2020 Aug 18;76(7):812-824. doi: 10.1016/j.jacc.2020.06.043. PMID 32792079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emergency care
Groups:
- Neuroprotect: MAP between 85-100mmHg SVO2 between 65-75%
  Neuroprotective goal directed hemodynamic optimization
Period: Overall Study
Arm/Group | Neuroprotect | Control
Started | 56 | 56
Completed | 52 | 55
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuroprotect | Control | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 65 (13) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 39 | 42 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 52 | 55 | 107

OUTCOME MEASURES:

1. Primary Outcome: % of Ischaemic Voxels With an ADC<0.65 mm2/s on Day 4-5 (Diffusion Weighted MRI)
Description: cerebral ischemia in post-cardiac arrest (CA) patients as quantified by the apparent diffusion coefficient (ADC) on diffusion weighted MRI (DW-MRI) to be performed at day 4- 5 post-CA using ADC scores in 11 pre-specified brain regions (frontal cortex, parietal cortex, temporal cortex, occipital cortex, precentral cortex, postcentral cortex, caudate nucleus, putamen, thalamus, cerebellum, pons).
Time Frame: day 4-5
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of ischaemic voxels
Arm/Group | Neuroprotect | Control
Number analyzed (Participants) | 52 | 55
percentage of ischaemic voxels | 10.6 [8.0 to 18.4] | 11.0 [8.4 to 14.8]
Statistical Analysis 1: Comparison: Control; missing data were accounted for by multiple imputation; Test type: Superiority; p = 0.0881, ANOVA; due to non normality of the residuals the data were log-transformed prior to the anova; Median ratio of final values = 1.37, 95% CI 2-sided [0.95 to 1.98] — the estimated mean difference obtained using the anova on the log-transformed data was back transformed thus yielding a ratio of median values

ADVERSE EVENTS:
Time Frame: During intervention period (36 hours)
Arm/Group | Neuroprotect | Control
All-Cause Mortality (participants affected / at risk) | 31/52 | 29/55
Serious Adverse Events (participants affected / at risk) | 7/52 | 21/55
Other Adverse Events (participants affected / at risk) | 0/52 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuroprotect (N=52) | Control (N=55)
arrhythmia (Cardiac disorders) | 7 (7) | 13 (13)
Limb ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
death (Cardiac disorders) | 0 (0) | 1 (1)
EMD (Cardiac disorders) | 1 (1) | 0 (0)
serious hypotension (Vascular disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02541591/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT02541591/SAP_001.pdf